#### APPENDIX II. WRITTEN INFORMED CONSENT DOCUMENT

## KEY INFORMATION FOR LONG-TERM HPV VACCINATION EFFECTIVENESS AND IMMUNITY IN RWANDAN WOMEN LIVING WITH OR WITHOUT HIV

We are asking you to choose whether or not to volunteer for a research study about how well the HPV vaccine works for women living in Rwanda. This page is designed to give you key information to help you decide whether to participate. We have included detailed information after this page. Ask the research team questions. If you have questions later, please contact the research investigator in charge of the study. Their contact information is below.

#### WHAT IS THE STUDY ABOUT AND HOW LONG WILL IT LAST?

Cancer of the cervix (the opening of the womb), anus, and throat can be caused by a virus – the human papillomavirus, also called HPV. We know that when the HPV vaccine is given to girls, it prevents infection from certain types of HPV. We want to understand how the vaccine prevents HPV infection for women many years after they were vaccinated. We also want to understand whether the vaccine works differently for women with HIV. By doing this study, we hope to learn among women like yourself in Rwanda, how well the vaccine works in the future. Your participation in this research will last about one year. Today, you will be asked to conduct a short questionnaire, provide a blood sample, and provide 3 samples of cells collected by a study nurse (vaginal, oral, and anal samples). If you do not have HIV, you will have an HIV test today. If any of these samples have HPV, we will ask you to return in 6-12 months for additional visits so you can provide samples again and see if you still have HPV or if it has gone away on its own. If you still have HPV, we may ask you to see a special doctor to make sure you do not have precancer.

#### REASONS YOU MIGHT CHOOSE TO VOLUNTEER FOR THIS STUDY

You will be adding to the knowledge of how HPV vaccination works in the future for women with different health conditions in Rwanda. Your participation will specifically help us understand how to improve HPV vaccination for women who live with HIV. For a complete description of benefits, refer to the Consent Document below.

#### REASONS YOU MIGHT CHOOSE NOT TO VOLUNTEER FOR THIS STUDY

We do not anticipate any mental, emotional, or physical harm through participation in this study. However, you may feel concerned about the confidentiality of the information shared as part of this research. Your responses will be kept completely confidential. None of the information you provide will be shared with anyone outside of the study team.

#### DO YOU HAVE TO TAKE PART IN THE STUDY?

Your participation is voluntary. You are being asked to complete the survey, but you may choose not to do so. You may choose to skip any questions that you do not wish to answer. If you sign the consent form document below, you have agreed to become part of the research study.

If you decide to take part, you are free to stop participating at any time without giving a reason. However, some of the information may have already been entered into the study and that will not be removed. The researchers may continue to use and share the information they have already collected.

## WHAT IF YOU HAVE QUESTIONS, SUGGESTIONS OR CONCERNS?

The person in charge of the study is Gad Murenzi, MD, MPH. If you have questions, suggestions, or concerns regarding this study or you want to withdraw from the study. His contact information is:

Gad Murenzi MD, MPH, Principal Investigator RD Rwanda, Kigali, Rwanda Tel: +250 788 589 085 / Email: gadcollins@gmail.com

If you are unable to reach Dr. Murenzi, Dr. Fabienne Shumbusho, MD is another researcher responsible for this study that you can reach out to. Her contact information is:

Dr. Fabienne Shumbusho, MD RD Rwanda, Kigali, Rwanda

Tel: +250 788 559 065 / Email: fabienneshumbusho@gmail.com

As the study will be conducted in Rwanda, if you wish to ask questions about the study or your rights as a research participant to someone other than the researchers or if you wish to voice any problems or concerns you may have about the study, please contact the chairperson of the Rwanda National Ethics Committee (RNEC) Dr. Mazarati Jean Baptiste at (250) 78830987 or Dr. Tumusiime David at (250) 788749398 or by mail: info@rnecrwanda.org.

If you have any additional questions, suggestions, or concerns about your rights as a volunteer in this research, contact staff in the Einstein Institutional Review Board (IRB) at <a href="irb@einstein.yu.edu">irb@einstein.yu.edu</a>.



# RWANDA NATIONAL ETHICS COMMITTEE/ALBERT EINSTEIN COLLEGE OF MEDICINE

## <u>DOCUMENTATION OF INFORMED CONSENT AND HEALTH INSURANCE</u> <u>PORTABILITY AND ACCOUNTABILITY ACT OF 1996 (HIPAA) AUTHORIZATION</u>

#### **Introduction**

You are being asked to participate in a research study called "Long-Term HPV Vaccination Effectiveness and Immunity in Rwandan Women Living with and without HIV". Your participation is voluntary -- it is up to you whether you would like to participate. It is fine to say "no" now or at any time after you have started the study. If you say "no," your decision will not affect any of your rights or benefits or your access to care.

Before you decide to be part of this research study, you need to understand the risks and benefits so that you can make an informed decision. This is known as informed consent. This consent form provides information about the study, which will also be explained to you. Once you understand the study and the risks involved, you will be asked to sign this form, or in the case that you are illiterate, provide your thumbprint on it and have it signed by a witness, if you want to take part. Remember, it is your decision: participation in the study is entirely voluntary.

If you cannot read, a study staff will help you read and understand the written paper that you will sign or thumbprint in the presence of a witness you trust, should you decide to join the study.

The researcher in charge of this project is called the "Principal Investigator." His name is **Gad Murenzi**, **MD**, **MPH**. You can reach Dr. **Murenzi** by phone at (250) 788589085. **Fabienne Shumbusho**, **MD** will be serving as a **Co-Investigator** of this study, and she can be reached by phone at (250) 0788559065. They are both researchers at:

Research for Development (RD Rwanda) and Rwanda Military Hospital

#### Kigali, Rwanda

For questions about the research study, or if you believe you have an injury, contact the Principal Investigator, Co-Investigator, RNEC or the Einstein IRB.

Support for this research study is provided by **the National Institutes of Health** (USA) through Grant No: 6U54CA190163-06.

The Rwanda National Ethics Committee (RNEC) and Institutional Review Board (IRB) of the Albert Einstein College of Medicine have approved this research study. The IRB # is in the stamp in the upper right-hand corner and bottom right corner as well.

If you have questions regarding your rights as a research subject, you may contact RNEC chairpersons **Dr. Mazarati Jean** Baptiste at (250) 78830987 or **Dr. Tumusiime David** at (250) 788749398. You can also reach the RNEC by email at <a href="mailto:info@rnecrwanda.org">info@rnecrwanda.org</a> or by mail:

Rwanda National Ethics Committee Ministry of Health P.O.Box.84 Kigali, Rwanda

If you have any additional questions, please feel free to contact the Einstein IRB at <a href="mailto:irb@einstein.yu.edu">irb@einstein.yu.edu</a>.

## Why is this study being done?

HPV infection is responsible for most of cancer of the cervix (the opening of the womb), especially for those women with HIV infection. Some other less-common cancers found in the anus and the throat are also caused by HPV. For over 10 years, a vaccine for HPV has been given to older girls in Rwanda. We know that when the HPV vaccine is given to girls, it prevents infection from certain types of HPV. We want to understand how the vaccine prevents HPV infection for women many years after they were vaccinated. We also want to understand whether the vaccine works differently for women with HIV. By doing this study, we hope to answer these questions.

#### Why am I being asked to participate?

You are being asked to take part in this study because you are a woman, aged 18-28 years of age, physically and mentally able and willing to participate in the study, and able and willing to provide written, informed consent, or else consent with a thumbprint.

#### What will happen if I participate in the study?

Today, in a private location at the study clinic you will complete a short questionnaire about your life, your reproductive health, and your sexual history. All your answers are strictly confidential. You do not have to respond to any question that makes you uncomfortable. You will provide a urine sample for a pregnancy test to confirm you are not pregnant. If you do not have HIV, you will take a rapid HIV test with a finger prick. A study nurse will provide counseling for you to understand what the results mean for you. A study nurse will collect a sample of your blood into a collection tube for testing on how your body responds to the HPV vaccine and possible infection. In a private exam room, the study nurse will help you swish a saline solution in your mouth and then spit it into a container. To collect cells from your vagina, the study nurse will insert a soft brush into your vagina, turn it three times and remove it. To collect cells from your anal canal the study nurse will insert a small swab into your anal canal, turn it for 20 seconds and remove it. Both collections are quick procedures with minimal discomfort. If all three samples do not have HPV, you are done with the study visits. If any of these three samples has HPV, we will ask you to return in 6-12 months for another visit so you can provide samples again and see if you still have HPV or if it has gone away on its own. If you still have HPV, we may ask you to see a special doctor to make sure you do not have precancer. At your visit with the special doctor, they will take one or more digital pictures of your cervix with a digital camera. The picture will not show the outside of your body, just the inside where the cervix is. Please note that the pictures will not identify you, and that picture of a cervix will not show your face or genitals. People cannot tell the specific woman from whom the cervix picture is taken. All pictures will be shown to you at the time if you want to see them.

#### How many people will take part in the research study?

You will be one of approximately 3,028 women participating in this study. We will be enrolling **1,514** women living with HIV and **1,514** women who are not infected with HIV.

#### Will there be audio and/or video recording?

No, there will be no audio or video recording in this study. You will hear an audio recording for the questionnaire that will be completed in private.

## **Information Banking (Future Use and Storage)**

- No testing of human genes will be conducted as part of the current study.
- ADDITIONAL TESTS ON YOUR SAMPLE: No other tests other than those explained under this study are currently planned.

However, if you agree, the specimens you provide for this research may be stored for future research testing. The specimen cannot be linked to you. In the future, researchers can apply for permission to use the specimen for new studies to prevent, diagnose or treat disease. Future testing may require samples to be analyzed in Rwanda, the United States, or elsewhere for testing. Your specimens/data may be kept for a long time, perhaps longer than 50 years.

If you agree to the future use, some of your de-identified specimens, digital pictures of your cervix and health information (not linked to you) may be placed into one or more scientific databases. Your specimens may also be submitted to a tissue/cell/DNA bank. You have the right to withdraw consent to use of the tissue for future use at any time by contacting the study doctors listed above. If that is your request, your unused specimens will be destroyed at the end of this study. Some researchers may develop tests, treatments or products that are worth money. You will not receive payment of any kind for your specimens/data or for any tests, treatments, products, or other things of value that may result from the research.

You can choose not to participate in the tissue/cell/DNA bank and still be part of the main study and this will not affect your treatment at this facility.

## PLEASE INDICATE YOUR CHOICE BY INITIALING ONE (1) OF THE FOLLOWING OPTIONS FOR EACH QUESTION

| 1. Specimens |
|---|
| I consent to have my specimens stored and used for future research studies. |
| I do NOT consent to have my specimens stored and used for future research studies. The |
| specimens will be destroyed at the end of the study. |
| 2. Future Contact About This Study |
| I consent to be contacted with general information about this study's research findings. |
| I do NOT consent to be contacted with general information about this study's research |
| indings. |
| 3. Future Research |
| I consent to being contacted about future research opportunities. |
| I do NOT consent to being contacted about future research opportunities. |

## Will I be compensated for being in this research study?

You will receive a total of 10,000 RWF in cash to compensate for your time and transport costs during the study visit and other follow-up visits if necessary. If you choose to withdraw from the study before all components of your participation are completed, you will be compensated only for the components you completed.

#### Will it cost me anything to participate in this study?

There will be no cost to you to participate in the study.

## **Confidentiality**

The researchers and study staff follow US federal, US state, and Rwandan laws to protect your privacy. This part of the consent form tells you what information about you may be used and shared in the research described in this form. You do not have to sign this form but, if you do not, you may not participate in the research.

The health information that we may use or disclose for the research described in this form includes information from your entire medical record, such as your name, phone number, email, medical diagnoses, dates, test results, social security number, medical record numbers, etc. In addition, the researchers wish to review information from your medical records pertaining to your HIV status and previous clinical care. If you are living with HIV or test positive for HIV today, the study staff may review information about your current and previous HIV care and laboratory tests from the health clinic. By law, you must specifically authorize access to these records:

| $\square$ Yes, I authorize the use an status. | d disclosure of my information pertaining to HIV testing and HIV |
|---|---|
| Initial: | Date: |

Your information and research records will be kept confidential. Your study information will be kept if they are useful for the research described in this form. The only people who can see your research records are:

- Researchers and other individuals who work with the researchers
- Organizations and institutions involved in this research, including those that fund the research, if applicable
- Groups that review research such as central reviewers, Institutional Review Boards, the Office for Human Research Protections, the US Food and Drug Administration, data coordinating centers, and domestic and foreign agencies that regulate research.

The purposes of these uses and disclosures are to (1) conduct the study and (2) make sure the study is being done correctly. The information covered under this form may no longer be protected by federal privacy laws (such as HIPAA) once disclosed, and those persons who receive your health information may share your information with others without your additional permission. All these groups are required to keep your information confidential.

#### **Certificate of Confidentiality**

As a way to protect your privacy, we have obtained a Certificate of Confidentiality from the National Institutes of Health, which is funding this study. If information from this study were requested or subpoenaed by government agencies or the courts, we would use the Certificate to attempt to legally refuse to provide that information. These requests are rare – in only a few cases did researchers have to use the Certificate, and it was honored most of the time, but not every time. There are several kinds of situations to which the Certificate does not apply. For example, we are still required to report child abuse and some diseases, and we must make data available to the government for review or evaluation of our research. The Certificate does not prevent you or a member of your family from voluntarily sharing information. Similarly, if an

insurer, employer, or other person obtains your written consent to receive research information, then the researchers may not use the Certificate to withhold that information.

## Are there any risks to me?

We do not think there are any physical risks related to participating in this research study. We will ask you questions about your sexual history and reproductive health that might make you feel uncomfortable. You have a right **not** to respond to any question that makes you uncomfortable.

A risk of taking part in this study is the possibility of a loss of confidentiality or privacy. Loss of privacy means having your personal information shared with someone who is not on the study team and was not supposed to see or know about your information. The study team plans to protect your privacy – see the Confidentiality section above for details.

However, there is occasionally the possibility of discomfort, bleeding, or bruising from the blood draw. These risks will be minimized by having a trained and experienced health worker draw your blood.

## Are there possible benefits to me?

Unless you are known to have HIV, you will have a rapid test and learn whether you have HIV. It is very unlikely that you have cervical or anal precancer. By participating in this study, any precancer diagnosed would be treated. More likely, you will not experience any direct benefit personally from participating in this study. We hope you will participate because the study will generate important information contributing to the knowledge of HPV vaccine effectiveness and immunity in Rwanda women living with or without HIV. Your participation will help to inform the development of programs and interventions for communities of people like yourself.

#### Will I get to know the results from this study?

If you have an HIV test, you will learn those results immediately. The result of the HPV infection test performed on you will not be communicated directly to you. However, if any of the three samples become positive, you may be contacted for follow-up visits approximately sixtwelve months later. And if, at follow-up visits, the HPV results remain positive, the study team may perform further tests to rule out precancer or refer you to the nearest specialized health service if there is any advanced disease. Some other results, which are obtained for research purposes only, will not be directly returned to you. However, the overall results of the research study will be made available to the public.

#### What choices do I have other than participating in this study?

You can refuse to participate in the study. If you decide not to participate, the medical care providers at this facility will still give you all standard care and treatment that is recommended for you.

#### Are there any consequences to me if I decide to stop participating in this study?

No. If you decide to take part, you are free to stop participating at any time without giving a reason. This will not affect your care and you will continue to be treated at this facility. However, some of the information may have already been entered into the study and that will not be removed. The researchers and the sponsor may continue to use and share the information they have already collected.

To withdraw your consent and authorization, you must contact the Principal or Co-Investigator in writing at the address on page 1 of this form. However, you may first call or speak to the Principal or co-Investigator and he/she will stop collecting new information about you. If you take back your consent and authorization, you will not be allowed to continue to participate in this research study.

## Who can answer my questions about the study?

You can talk to the research team member that explains the study to you about any questions, concerns, or complaints. You may also telephone Dr. Gad Murenzi / Dr. Fabienne Shumbusho on 0788589085/0788559065. If you wish to ask questions about the study or your rights as a research participant to someone other than the researchers or if you wish to voice any y

| Tights we will be with purity to be middle control than the labell that of it job with the vertex will |
|---|
| problems or concerns you may have about the study, please contact: RNEC chairperson <b>Dr.</b> |
| Mazarati Jean Baptiste at (250) 78830987 or Dr. Tumusiime David at (250) 788749398 or b |
| mail: info@rnecrwanda.org |
| Consent |
| You have been given a copy of this consent form. |

Declaration

## **CONSENT TO PARTICIPATE**

I have read the consent form and I understand that it is up to me whether I participate. I know enough about the purpose, methods, risks, and benefits of the research study to decide that I want to take part in it. I understand that I am not waiving any of my legal rights by signing this informed consent document. I will be given a signed copy of this consent form.

| Printed name of participant | Signature or thumbprint of participant | Date |
|---|---|---|
| Printed name of the person conducting the consent process | Signature | Date |

If the person is unable to read and/or write, an impartial witness should be present during the informed consent discussion. After the informed consent form is read and explained to the person, and after they have orally consented to their participation in the study and have either signed the consent form or provided their fingerprint, the witness should sign and personally date the consent form. By signing the consent form, the witness attests that the information in the consent form and any other written information was accurately explained to, and apparently understood by, the person and that informed consent was freely given by the person.

| Printed name of witness if participant utilized a thumbprint to consent to participation in this study | Signature of witness | Date |
|---|---|---|
| | | _ |
| Printed name of the person conducting the | Signature | Date |